CLINICAL TRIAL: NCT03285204
Title: Relationship Between Neurological Disability and Visual Impairment in Patients With ALS or Friedreich's Ataxia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Jose Luis Urcelay Segura (Other)
Responsible Party: Sponsor-Investigator, Jose Luis Urcelay Segura, Head Of ophthalmology, Hospital General Universitario Gregorio Marañon
Organization: Hospital General Universitario Gregorio Marañon (Other)
Other Study IDs: ELA-AF-OCT-2014-01
Record Dates: First submitted 2017-03-08; First posted 2017-09-15 (Actual); Last update posted 2019-02-26 (Actual); Status verified 2018-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: optical coherence tomography; amyotrophic lateral sclerosis
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- ALS patients
- Friedreich Ataxia patients
- Healthy control

SUMMARY:
The aim of this study is to obtain an early biomarker of amyotrophic lateral sclerosis and Friedreich's Ataxia which allows to diagnose the disease in an initial stage and to follow up the patient with optic coherence tomography, a fast, non-invasive and comfortable method

DETAILED DESCRIPTION:
All patients will be asked about their data and their general medical history, and will be underwent on one hand, a complete neurological examination including the degree of neurological impairment quantified according to the functional rating scale of ALS (ALSFRS-r) or Scale for the assessment and rating of ataxia (SARA); On the other hand, they will have a complete ophthalmological examination too, including the patient's graduation, pupillary and ocular motility examination, biomicroscopy, Goldman tonometry and fundus exam. Patients will be performed too a conventional automated Humprey perimetry, color test (Farnsworth-Munsell 28 Hue Color Vision Test) and finally an optical coherence tomography (OCT) in order to see possible anatomical alterations in both macula and optic nerve. The follow-up of these explorations will be repeated in all cases at 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years.
* Best corrected visual acuity more than 0.4 (20/50 Snellen = 0.4 logMAR = 65 ETDRS letters).
* Refractive defect less than 5 diopters of spherical equivalent and / or cylinder less than 2 diopters.
* Transparent optical media: Opacity of crystalline <1 according to Lens Opacities Classification System (LOCS) III.
* Open anterior chamber angle assessed by gonioscopy with Goldmann lens (grade> III).
* Availability and collaboration to carry out the tests of the exploratory protocol.
* Acceptance of informed consent.

Exclusion Criteria:

* Previous intraocular surgeries of less than 6 months of evolution. Patients with refractive surgery using the LASIK or LASEK technique will not be excluded.
* Physical or mental difficulties to perform reliable and reproducible perimeters.
* Pathology and / or ocular malformations, angular or optic nerve anomalies.
* Any retinopathy or maculopathy.
* Intraocular pressure (IOP)> 21 mmHg.
* Signal-to-noise ratio in OCT less than 5/10.
* Failure to meet any inclusion criteria.
* Mental retardation or any other limitation in obtaining informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Amyotrophic lateral sclerosis patients Friedreich's ataxia patients Healthy volunteers
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2015-07 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2020-02 (Estimated)

PRIMARY OUTCOMES:
early biomarker of amyotrophic lateral sclerosis and Friedreich's Ataxia | change from baseline to 6 month
  macular, ganglion cell layer and retinal nerve fiber layer thickness measure

CONTACTS AND LOCATIONS:
Overall Officials: Jose L Urcelay, PhD, Principal Investigator — HGU Gregorio Marañón
Locations (1):
- Pilar Rojas Lozano, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No